CLINICAL TRIAL: NCT05286801
Title: A Phase 1/2 Study of Tiragolumab (NSC# 827799) and Atezolizumab (NSC# 783608) in Patients With Relapsed or Refractory SMARCB1 or SMARCA4 Deficient Tumors
Brief Title: Tiragolumab and Atezolizumab for the Treatment of Relapsed or Refractory SMARCB1 or SMARCA4 Deficient Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-01992; NCI-2022-01992 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2121 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2121 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Atypical Teratoid/Rhabdoid Tumor; Epithelioid Sarcoma; Kidney Medullary Carcinoma; Malignant Solid Neoplasm; Poorly Differentiated Chordoma; Recurrent Atypical Teratoid/Rhabdoid Tumor; Recurrent Chordoma; Recurrent Epithelioid Sarcoma; Recurrent Kidney Medullary Carcinoma; Recurrent Malignant Solid Neoplasm; Recurrent Rhabdoid Tumor; Refractory Atypical Teratoid/Rhabdoid Tumor; Refractory Chordoma; Refractory Epithelioid Sarcoma; Refractory Kidney Medullary Carcinoma; Refractory Malignant Solid Neoplasm; Refractory Rhabdoid Tumor; Rhabdoid Tumor
MeSH Terms: conditions — Rhabdoid Tumor; Sarcoma; Chordoma | interventions — atezolizumab; Specimen Handling; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Tiragolumab; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B (atezolizumab, tiragolumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1 and tiragolumab IV over 30-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients also undergo standard imaging scans including x-rays, CT, MRI, and/or FDG PET-CT throughout the trial. Patients also undergo ECHO during screening and blood sample collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tiragolumab; Procedure: X-Ray Imaging
- Part A (atezolizumab, tiragolumab) (Experimental): Patients receive tiragolumab IV over 30-90 minutes on day 1 of each cycle and atezolizumab IV over 30-60 minutes on day 1 of each cycle starting in cycle 2. Treatment repeats every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo standard imaging scans including x-rays, CT, MRI, and/or FDG PET-CT, throughout the trial. Patients also undergo ECHO during screening and blood sample collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tiragolumab; Procedure: X-Ray Imaging

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT and/or PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Part A (atezolizumab, tiragolumab)
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET-CT and/or FDG-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Tiragolumab — Given IV
  Other Names: MTIG7192A; RG6058
Procedure: X-Ray Imaging — Undergo x-rays
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase I/II trial studies how well tiragolumab and atezolizumab works when given to children and adults with SMARCB1 or SMARCA4 deficient tumors that have either come back (relapsed) or do not respond to therapy (refractory). SMARCB1 or SMARCA4 deficiency means that tumor cells are missing the SMARCB1 and SMARCA4 genes, seen with some aggressive cancers that are typically hard to treat. Immunotherapy with monoclonal antibodies, such as tiragolumab and atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of tiragolumab as monotherapy in pediatric patients (< 18 years) with SMARCB1 or SMARCA4 deficient tumors. (Part A) II. To evaluate antitumor activity of the combination of tiragolumab and atezolizumab as assessed by objective response rate in patients with SMARCB1 or SMARCA4 deficient tumors per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 (for non-central nervous system [CNS] tumors) or CNS response criteria (for CNS tumors). (Part B) III. To evaluate the safety and adverse event profile of this combination therapy in subjects with SMARCB1 or SMARCA4 deficient tumors, with a particular focus in pediatric patients < 12 years of age.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of tiragolumab alone in part A and tiragolumab and atezolizumab (part A and B) when given in combination in pediatric, AYA (adolescents and young adults), and adult patients.

II. To estimate the PFS (progression free survival), OS (overall survival), and duration of response of combination tiragolumab and atezolizumab in patients with SMARCB1 or SMARCA4 deficient tumors.

EXPLORATORY OBJECTIVES:

I. To evaluate molecular features of the SMARCB1 or SMARCA4 tumors including genomic and transcriptomic evaluation and if feasible, assess their association to clinical response.

II. To assess the association of response rate to the molecular subtypes of rhabdoid/atypical teratoid rhabdoid tumor (ATRT).

III. To assess changes in circulating and tumoral immune markers in patients treated with this combination therapy and correlate to response when feasible.

OUTLINE: Patients are assigned to Part A or Part B.

PART A: Patients receive tiragolumab intravenously (IV) over 30-90 minutes on day 1 of each cycle and atezolizumab IV over 30-60 minutes on day 1 of each cycle starting in cycle 2. Treatment repeats every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo standard imaging scans including x-rays, computed tomography (CT), magnetic resonance imaging (MRI), and/or positron emission tomography (PET)-CT throughout the trial. Patients also undergo echocardiography (ECHO) during screening and blood sample collection on study.

PART B: Patients receive atezolizumab IV over 30-60 minutes on day 1 and tiragolumab IV over 30-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients also undergo standard imaging scans including x-rays, CT, MRI, and/or FDG PET-CT, throughout the trial. Patients also undergo ECHO during screening and blood sample collection on study.

After completion of study treatment, patients are followed up at months 3, 6, 9, 12, 18, 24, 36, 48, and 60, up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 12 months of age at the time of study enrollment. For part A, patients must be < 18 years old at enrollment. For part B, there is no upper age limit

  * The Part B (phase 2) cohorts will initially open concurrently with the part A but will only enroll patients at least 18 years of age. Patients < 18 years of age will be included in the part B cohorts only after the tiragolumab monotherapy dose has been assessed to be safe in the part A portion
* Patients must have SMARCB1 (INI1) or SMARCA4 deficient tumors verified through institutional immunohistochemistry (IHC) or molecular confirmation of a pathologic SMARCB1 (INI1) or SMARCA4 loss or mutation in the tumor from a Clinical Laboratory Improvement Act (CLIA) certified lab with the following disease histologies:

  * Renal medullary carcinoma
  * Malignant rhabdoid tumor (extra-CNS)
  * Atypical teratoid rhabdoid tumor (CNS)
  * Poorly differentiated chordoma
  * Epithelioid sarcoma
  * Other SMARCB1 or SMARCA4 deficient tumors
  * Note: Molecular studies will only be used if IHC is equivocal or cannot be performed. Documentation of the institutional IHC or molecular testing must be uploaded via the RAVE system
* Part A: Patients must have either measurable or evaluable disease Part B: Patients must have measurable disease per RECIST v1.1 for non-CNS tumors or CNS response criteria for CNS tumors

  * Note: See protocol for specific exclusion for patients with CNS primary or metastatic disease
* Patients must have relapsed, refractory disease or newly diagnosed disease for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2 (Karnofsky/Lansky score of >= 50). Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: See Developmental Therapeutics (DVL) homepage on the Children's Oncology Group (COG) Members site for commercial and investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment

    * >= 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea). Please refer to the table of myelosuppressive/Anticancer Agents on the COG website: https://www.cogmembers.org/uploadedFiles/Site/Disc/DVL/Documents/TableOfMyelosuppressiveAnti-CancerAgents.pdf
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent. See the DVL homepage on the COG Members site for commercial and investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total-body irradiation [TBI]):

    * Autologous stem cell infusion including boost infusion: >= 30 days
  * Cellular therapy: >= 30 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * External radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 90 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iodine I 131 metaiodobenzylguanidine [131I MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have had prior TIGIT targeting therapy
  * Patients must not have received prior therapy with an anti- PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA4 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (i.e. OX-40, CD137)
  * Patients must not have received live/attenuated vaccine within 30 days of first dose of treatment
  * Patients must not be receiving concomitant systemic steroid medications and >= 14 days must have elapsed since last dose of systemic corticosteroid with the following exceptions:

    * The use of physiologic doses of corticosteroids (5 mg/m^2/day up to 10 mg/day of prednisone equivalent) is acceptable
    * The use of topical, inhaled, or ophthalmic corticosteroids are acceptable
    * The use of acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are acceptable
  * Treatment with systemic immunosuppressive medication (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha [TNF-alpha] agents) must have concluded >= 14 days prior to study enrollment
* For patients with solid tumors without known bone marrow involvement

  * Peripheral absolute neutrophil count (ANC) >= 1000/uL (must be performed within 7 days prior to enrollment)
* For patients with solid tumors without known bone marrow involvement

  * Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (must be performed within 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts above (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity
* A creatinine based on age/sex as follows (must be performed within 7 days prior to enrollment):

  * Age; Maximum Serum Creatinine (mg/dL)

    * 1 to < 2 years; Male: 0.6; Female: 0.6
    * 2 to < 6 years; Male: 0.8; Female: 0.8
    * 6 to < 10 years; Male: 1; Female: 1
    * 10 to < 13 years; Male: 1.2; Female: 1.2
    * 13 to < 16 years; Male: 1.5; Female: 1.4
    * >= 16 years; Male: 1.7; Female: 1.4 OR- a 24 hour urine creatinine clearance >= 70 mL/min/1.73 m^2 (must be performed within 7 days prior to enrollment) OR- a glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard) (must be performed within 7 days prior to enrollment)
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Bilirubin (sum of conjugated + unconjugated or total) =< 1.5 x upper limit of normal (ULN) for age (must be performed within 7 days prior to enrollment)

  * Patients with known Gilbert disease: Total bilirubin =< 3 x ULN
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (must be performed within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L
* Albumin >= 2 g/dL (must be performed within 7 days prior to enrollment)
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] v5) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible
* International normalized ratio (INR) =< 1.5 (must be performed within 7 days prior to enrollment)
* Serum amylase =< 1.5 x ULN (must be performed within 7 days prior to enrollment)
* Serum lipase =< 1.5 x ULN (must be performed within 7 days prior to enrollment)
* Grade 1 or lower calcium level

  * Note: can have history of hypercalcemia as long as controlled and asymptomatic

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in female patients of childbearing potential. Female patients of childbearing potential are defined as those who are past the onset of menarche and are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, complete hysterectomy) or post-menopausal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of therapy and at least 90 days after final dose of tiragolumab and 150 days after final dose of atezolizumab, whichever is later. Abstinence is an acceptable method of birth control.

  * It is not known if atezolizumab or tiragolumab are present in breast milk; however, IgG immunoglobulins are found in milk. Due to the potential for serious adverse reactions in the breastfed infant, breastfeeding is not recommended during therapy and for at least 150 days after the last dose of atezolizumab and 90 days after the last dose of tiragolumab, whichever is later
* Concomitant medications:

  * Corticosteroids:

    * Patients must not be receiving concomitant systemic steroid medications and >= 14 days must have elapsed since last dose of systemic corticosteroid with the following exceptions:

      * The use of physiologic doses of corticosteroids (5 mg/m^2/day up to 10 mg/day of prednisone equivalent) is acceptable
      * The use of topical, inhaled, or ophthalmic corticosteroids are acceptable
      * The use of acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g. 48 hours of corticosteroids for a contrast allergy) are acceptable
  * Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible
  * Systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, and thalidomide) during study treatment because these agents could potentially alter the efficacy and safety of study treatments would not be eligible
* Patients must not have a known hypersensitivity to any component of tiragolumab or atezolizumab injection
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation
* Patients who have undergone allogeneic bone marrow or allogeneic cell transplant are not eligible
* Patients with CNS metastases from non-CNS primary tumors are not eligible unless CNS metastases have been previously treated and sequential imaging shows no evidence for active disease in the CNS.

  * Patients with primary CNS tumors (including ATRT) with involvement of the brainstem are not eligible. Note: Patients with ATRT with M0-M4 disease without involvement of the brain stem are allowed to participate
* Patients must not have active autoimmune disease that has required systemic treatment in the past 12 months, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are not excluded. Replacement therapy (e.g. thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and these patients are eligible
* Patients who have active immune deficiency are not eligible
* Patients who have known active tuberculosis are not eligible
* Hepatitis B or C infection:
* Patients < 18 years old at enrollment, who have known hepatitis B or C
* Patients >= 18 years old at enrollment with:

  * Positive hepatitis B surface antigen (HBsAg), OR
  * Positive total hepatitis B core antibody (HBcAb) who have a quantitative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) >= 500 IU/mL, OR
  * Positive hepatitis C virus (HCV) antibody with a positive HCV ribonucleic acid (RNA) test
  * Note: For adults (>= 18 years old at enrollment), hepatitis B serology testing is required to determine eligibility. The HBV DNA test is required only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test. For adults (>= 18 years old at enrollment), hepatitis C serology testing is required to determine eligibility. The HCV RNA test is required only for patients who have a positive HCV antibody test
* Patients who have a known, recent Epstein-Barr virus (EBV) infection or known history of chronic, active infection are not eligible
* Patients who have history of or active human immunodeficiency virus (HIV) are not eligible except patients who are stable on anti-retroviral therapy, have a CD4 count >= 200/uL, and have an undetectable viral load
* Patients who have significant cardiovascular disease (such as New York Heart Association class III or IV congestive heart failure, myocardial infarction, or cerebrovascular accident) within 3 months prior to study enrollment, unstable arrhythmia, or unstable angina are not eligible
* Patients who have a major surgical procedure, other than for diagnosis, within 4 weeks prior to study enrollment, or the anticipation of the need for a major surgical procedure during the study are not eligible
* Patients who have a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or known active pneumonitis are not eligible. History of radiation pneumonitis in the radiation field is permitted
* Patients who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) are not eligible. Patients with indwelling catheters (e.g., PleurX) are allowed
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of cycle 1 dose limiting toxicities of tiragolumab as monotherapy in pediatric patients | Up to 21 days
  Frequency (%) of pediatric patients (<18 years) with cycle 1 dose limiting toxicities attributable to tiragolumab as monotherapy in the safety cohort (Part A).
Frequency of objective response for the combination of tiragolumab and atezolizumab | Up to 5 years
  Frequency (%) of patients with best objective response of partial or complete for the combination of tiragolumab and atezolizumab stratified by disease cohort (Part B).
Frequency of cycle 1 dose limiting toxicities of the combination of tiragolumab and atezolizumab in patients < 12 years | Up to 21 days
  Frequency (%) of patients < 12 years with cycle 1 dose limiting toxicities attributable to the combination of tiragolumab and atezolizumab in Part B.

SECONDARY OUTCOMES:
Trough concentration of tiragolumab as monotherapy in cycle 1 | Up to 21 days
  Median (min, max) of trough concentration for tiragolumab as monotherapy in cycle 1 of Part A safety cohort patients (< 18 years).
Trough concentration for tiragolumab when given in combination with atezolizumab in cycle 2, day 1 | Up to 21 days
  Median (min, max) of trough concentration for tiragolumab when given in combination with atezolizumab in cycle 2, day 1 of Part B cohorts stratified by age group (< 18 versus >= 18 years) and disease cohort.
Trough concentration for atezolizumab when given in combination tiragolumab with in cycle 3, day 1 | Up to 21 days
  Median (min, max) of trough concentration for atezolizumab when given in combination tiragolumab in cycle 3, day 1 of Part B cohorts stratified by age group (< 18 versus >= 18 years) and disease cohort.
Progression free survival (PFS) of the combination therapy for tiragolumab and atezolizumab | Up to 5 years
  Median (95% CI) progression-free survival for the combination therapy of tiragolumab and atezolizumab stratified by disease cohort in Part B.
Overall survival (OS) of the combination therapy for tiragolumab and atezolizumab | Up to 5 years
  Median (95% CI) for the combination therapy of tiragolumab and atezolizumab stratified by disease cohort in Part B.
Duration of response of the combination therapy for tiragolumab and atezolizumab | Up to 5 years
  Median (min, max) duration of response among patients in Part B with partial or complete response to combination therapy for tiragolumab and atezolizumab stratified by disease cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Wedekind Malone, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (40):
- United States (35):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT05286801/ICF_000.pdf